CLINICAL TRIAL: NCT07177625
Title: Assessment of Patient Comfort and Analgesic Efficacy of Retrolaminar Block During Extracorporeal Shock Wave Lithotripsy : An Observational Prospective Study
Brief Title: Retrolaminar Block Analgesia and Patient Comfort During Prone ESWL
Status: Not yet recruiting | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Serpil Bayındır, Specialist Doctor, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: FSCH-SBÜ-2025/09
Record Dates: First submitted 2025-08-26; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Urolithiasis
Keywords: Extracorporeal Shock Wave Lithotripsy; Retrolaminar block; Prone position
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: RLB Group - Retrolaminar block prior to ESWL: Participants in this group will receive an ultrasound-guided retrolaminar block prior to prone-position ESWL. The block will be performed using [specify local anesthetic type and dose]. All ESWL procedures will be performed according to standard hospital protocols. Patients will be monitored for pain intensity (VAS), vital signs, procedural duration, and any adverse events during and after the procedure. Rescue analgesia will be administered if necessary.
  Interventions: Procedure: Retrolaminar block
- Sedation Group - Standard sedoanalgesia: Participants in this group will receive standard sedoanalgesia during prone-position ESWL using [specify drug(s), dose, and infusion method]. Pain intensity (VAS), vital signs, procedural duration, and any adverse events will be monitored throughout and after the procedure. Rescue analgesia will be provided as needed according to hospital protocols.
  Interventions: Drug: Sedoanalgesia
- Control Group - No additional block or sedoanalgesia: Participants in this group will undergo prone-position ESWL without any additional regional block or sedoanalgesia. Standard monitoring of pain intensity (VAS), vital signs, procedural duration, and any adverse events will be conducted. Rescue analgesia will be provided if clinically indicated.
  Interventions: Other: No Intervention / None

INTERVENTIONS:
Procedure: Retrolaminar block — Ultrasound-guided retrolaminar block performed prior to prone-position ESWL. This intervention is applied only to participants in the RLB Group. Patients will be monitored for pain intensity (VAS), vital signs, procedural duration, and any adverse events during and after the procedure. Rescue analgesia will be administered if clinically indicated.
  Other Names: RLB Group
  Groups: Group 1: RLB Group - Retrolaminar block prior to ESWL
Drug: Sedoanalgesia — Standard sedoanalgesia administered during prone-position ESWL. This intervention is applied only to participants in the Sedation Group. Pain intensity (VAS), vital signs, procedural duration, and any adverse events will be monitored. Rescue analgesia will be provided as needed.
  Groups: Sedation Group - Standard sedoanalgesia
Other: No Intervention / None — No additional regional block or sedoanalgesia; standard monitoring only. This applies only to participants in the Control Group. Pain intensity (VAS), vital signs, procedural duration, and any adverse events will be monitored. Rescue analgesia will be provided if clinically indicated.
  Groups: Control Group - No additional block or sedoanalgesia

SUMMARY:
The purpose of this prospective, observational study is to evaluate the effect of retrolaminar block (RLB) on patient comfort and analgesic effectiveness during extracorporeal shock wave lithotripsy (ESWL) procedures. The main questions the study aims to answer are:

Does retrolaminar block reduce pain intensity during ESWL?

Does retrolaminar block improve patient comfort during ESWL?

Participants will undergo the following interventions:

RLB Group: Retrolaminar block performed under ultrasound guidance prior to ESWL.

Sedation Group (S): Standard sedoanalgesia administered.

Control Group (C): No additional regional block or sedoanalgesia applied.

Participants will be monitored for pain levels, procedural duration, hemodynamic parameters, and the need for additional analgesics. The study aims to determine whether retrolaminar block can serve as a safe and effective analgesic method during ESWL procedures.

DETAILED DESCRIPTION:
This prospective, observational study aims to investigate the effect of retrolaminar block (RLB) on analgesic efficacy and patient comfort during extracorporeal shock wave lithotripsy (ESWL). Adult patients scheduled for ESWL will be enrolled and allocated into three groups:

RLB Group: Retrolaminar block performed under ultrasound guidance prior to ESWL.

Sedation Group (S): Standard sedoanalgesia administered.

Control Group (C): No additional regional block or sedoanalgesia applied.

Pain intensity will be assessed using the Numeric Rating Scale (0-10) at multiple time points during and after the procedure. Procedural duration, hemodynamic parameters, and need for rescue analgesics will also be recorded. Patient comfort and satisfaction will be evaluated immediately post-procedure and at recovery. Safety outcomes, including adverse events related to RLB or sedoanalgesia, will be monitored.

The study seeks to determine whether retrolaminar block is a safe and effective analgesic technique for ESWL, potentially improving patient comfort while reducing systemic analgesic requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA Physical Status I-III
* Undergoing ESWL in prone position
* Provided written informed consent

Exclusion Criteria:

* ASA Physical Status IV or higher
* Allergy to local anesthetics or sedatives
* Coagulopathy or anticoagulant use
* Local infection at injection site
* Severe spinal deformity or anatomical abnormality preventing block
* Cognitive impairment or inability to use VAS
* Pregnancy
* Chronic opioid use or chronic pain medication
* Emergency ESWL
* Previous open surgery at block site
* Intraoperative hemodynamic instability or severe complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for ESWL for urinary system stones at Elazığ Fethi Sekin City Hospital. Participants will be assigned to receive Retrolaminar Block, standard sedoanalgesia, or no intervention. Pain intensity, vital signs, procedural parameters, and adverse events will be monitored.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Assessed using the Visual Analog Scale (VAS; 0 = no pain, 10 = worst pain) at four time points: baseline, immediately post-procedure, 30 minutes post-procedure, and 60 minutes post-procedure.
  Pain intensity will be assessed using the Visual Analog Scale (VAS; 0 = no pain, 10 = worst pain) at four time points: before ESWL (baseline), immediately after the procedure, 30 minutes post-procedure, and 60 minutes post-procedure. This outcome evaluates the analgesic effectiveness of Retrolaminar Block, Sedoanalgesia, or no intervention.

SECONDARY OUTCOMES:
Rescue Analgesia Requirement | During and up to 60 minutes post-procedure.
  The need for additional analgesia during and after ESWL will be recorded to evaluate differences between the groups (RLB, Sedoanalgesia, Control). Recorded as type, dose, and timing of additional analgesics
Heart rate | Throughout the ESWL procedure (from initiation until termination, typically 30-90 minutes), with measurements recorded every 10 minutes
  Heart rate will be monitored throughout the ESWL procedure and recovery period to assess hemodynamic stability.
Adverse Events | During procedure and up to 60 minutes post-procedure
  Any adverse events related to ESWL, sedation, or block will be documented.
Noninvasive Blood Pressure | Throughout the ESWL procedure (from initiation until termination, typically 30-90 minutes), with measurements recorded every 10 minutes
  Noninvasive Blood Pressure will be monitored to assess hemodynamic stability
Oxygen Saturation | Throughout the ESWL procedure (from initiation until termination, typically 30-90 minutes), with measurements recorded every 10 minutes
  Oxygen saturation will be monitored to ensure adequate oxygenation and patient safety throughout the procedure and recovery.
Global Assessment of Quality of Life (Physician's Global Assessment) | Within 1 hour after ESWL procedure
  Physicians will provide a global assessment of patient well-being using a 10-point numeric rating scale (0 = poorest outcome, 10 = best outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No